CLINICAL TRIAL: NCT03527680
Title: Effect of Lactobacillus Rhamnosus on Serum Uremic Toxins (Phenol and P-Cresol ) in Hemodialysis Patients: A Double Blind Randomized Clinical Trial
Brief Title: Effect of Lactobacillus Rhamnosus on Serum Uremic Toxins in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: nooshin dalili (Other)
Responsible Party: Sponsor-Investigator, nooshin dalili, assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRCT20154182017N21
Record Dates: First submitted 2017-05-21; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus rhamnosus (Experimental): received daily one capsule containing 1.6*107 CFU of Lactobacillus Rhamnosus
  Interventions: Dietary Supplement: Lactobacillus rhamnosus
- Placebo (Placebo Comparator): received one placebo capsule per day Infant formula after meal for 28 days
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus — daily one capsule containing 1.6*107 CFU of Lactobacillus Rhamnosus prepared by Tabriz Nutrition Research Center from yogurt and cheese of different farms located in the suburbs Heris, after meal for 28 days
  Arms: Lactobacillus rhamnosus
Drug: Placebo - Cap — daily one capsule of placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Uremic toxins such as p-cresol and phenol are suggested to be associated with higher mortality in hemodialysis patients. The aim of this study was to investigate the effects of probiotics on serum p-cresol level in hemodialysis patients.

DETAILED DESCRIPTION:
Overall, 42 hemodialysis patients (10 women and 32 men) were divided randomly into the Lactobacillus rhamnosus group (21 patients) and the placebo group (21 patients).

ELIGIBILITY:
Inclusion Criteria:• Age more than 20 years

* Acceptable performance of alimentary system
* Ability to drink at least 200 ml of water per day
* No history of being allergic to fungi and yeast
* Absence of acute medical illness
* life expectancy more than 3 months
* Accept and sign the consent

Exclusion Criteria:

* Patient's unwillingness to participate in the study
* History of smoking, peritoneal dialysis (PD) or previous kidney transplantation
* Lactation or pregnancy
* Drug history including antibiotics, prebiotics, probiotics, herbal drugs, psychedelic drugs, flavors.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
pre- and post-treatment p-cresol levels | 4 weeks

IPD SHARING:
Plan to Share IPD: Undecided